CLINICAL TRIAL: NCT06187662
Title: BrighT STAR LIBRA: Leveraging Implementation Science for Blood Culture Reduction Approaches
Acronym: LIBRA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 23-021013; 5K23HL151381-03 (NIH)
Record Dates: First submitted 2023-12-18; First posted 2024-01-02 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Blood Culture Rates; Antibiotic Stewardship; Implementation Science
Keywords: blood culture; antibiotic stewardship; implementation
MeSH Terms: interventions — Checklist

STUDY DESIGN:
Intervention Model Description: Study sites will be randomized into two arms, in which different strategies are introduced that each target distinct determinants of blood culture overuse
Who Masked: Participant, Care Provider
Masking Description: The primary study team will know which arm the participating site PICUs will be in, but the local study team and care teams will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Default Bias (Experimental): This intervention consists of a checklist to guide blood culture decisions, that a clinician in a site randomized to Arm A will be asked to consult and complete prior to ordering or not ordering a blood culture; as the relevant clinical scenario occurs.
  Interventions: Behavioral: Checklist
- Loss Aversion (Experimental): This intervention consists of targeted messaging and education that the primary study team will create and ask the Arm B sites to deliver to the PICU clinicians, which focuses on the importance of diagnostic stewardship and the current evidence for the benefit/low risk nature of the stewardship program to date.
  Sites in this arm will also receive a checklist to guide blood culture decisions, that clinicians at sites will be asked to consult and complete prior to ordering or not ordering a blood culture.
  Interventions: Behavioral: Checklist; Behavioral: Targeted Messaging

INTERVENTIONS:
Behavioral: Checklist — This intervention consists of a checklist to guide blood culture decisions, that a clinician in a site randomized to Arm A will be asked to consult and complete prior to ordering or not ordering a blood culture; as the relevant clinical scenario occurs. Meaning, if a clinician in Arm A is faced with a scenario in which it is customary or usual care to consider a blood culture, the clinician will be asked to first review this checklist. The checklist is not a binding or absolute process - the clinician should use both the checklist and typical clinical judgment to decide if the blood culture test is needed or not. The checklist is based on prototypes used in the completed parent study, BrighT STAR and the earlier preliminary studies at Johns Hopkins.
Behavioral: Targeted Messaging — This intervention consists of targeted messaging and education that the primary study team will create and ask the Arm B sites to deliver to the PICU clinicians, which focuses on the importance of diagnostic stewardship and the current evidence for the benefit/low risk nature of the stewardship program to date.
  Arms: Loss Aversion

SUMMARY:
This study will compare two strategies that target distinct determinants of blood culture overuse in an exploratory, hybrid, pilot trial in 8 PICUs. It aims to determine if there is any association between specific strategies used to reduce blood culture overuse on unit-wide blood culture rates, patient safety, and concurrently explore aspects of the implementation process (acceptability, feasibility, appropriateness).

DETAILED DESCRIPTION:
Blood cultures are an important test to diagnose bacterial bloodstream infections, but can be ordered reflexively, excessively, and lead to downstream negative patient consequences such as unnecessary antibiotic exposure. Work to date has demonstrated safe and effective reduction in blood culture rates in the pediatric intensive care unit (PICU) setting, but optimal strategies to reduce culture use are currently unknown.

The primary study team will initially work with all enrolled sites in an identical fashion, facilitating a core series of steps for implementing a quality improvement blood culture diagnostic stewardship program which is identical to the steps used in the parent study, called BrighT STAR (Testing STewardship to reduce Antibiotic use and Resistance). In addition, the primary study team will randomize sites into two arms, in which different strategies are introduced that each target distinct determinants of blood culture overuse. The primary study team will examine the impact on blood culture rates, as well as evaluate aspects of the implementation process, in all sites pre- vs-post intervention.

ELIGIBILITY:
Inclusion Criteria:

* Males or females over 18 years old
* PICU clinicians with direct patient care roles

Exclusion Criteria:

* Non-English speaking
* PICU clinicians who report to the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Total Blood Culture Rates | Approximately 24 months
  Compare differences in clinical outcomes, via total blood culture rates, before and after intervention, as well as between intervention arms
Acceptability of Intervention Measure (AIM) | one year
  Compare differences in implementation outcomes, via AIM surveys, before and after intervention, as well as between intervention arms. The AIM survey consists of a 4-item measure using a 5-point Likert scale, where 1=Completely disagree and 5=Completely agree
Intervention Appropriateness Measure | one year
  Compare differences in implementation outcomes, via Implementation Appropriateness Measure (IAM) surveys, before and after intervention, as well as between intervention arms. The IAM survey consists of a 4-item measure using a 5-point Likert scale, where 1=Completely disagree and 5=Completely agree
Feasibility of Intervention Measure (FIM) | one year
  Compare differences in implementation outcomes, via FIM surveys, before and after intervention, as well as between intervention arms. The FIM survey consists of a 4-item measure using a 5-point Likert scale, where 1=Completely disagree and 5=Completely agree

SECONDARY OUTCOMES:
Safety Outcomes Post-Intervention | one year
  Monitor safety outcomes of the blood culture diagnostic stewardship program in all sites, defined as episodes of delay in diagnosis of bacteremia in enrolled sites post-implementation of the pilot study; using chart review and a standardized safety event review form that is identical to the completed parent study, BrighT STAR.

OTHER OUTCOMES:
Qualitative Interview Data | one year
  Analyze qualitative interview data from each sites' lead team members to better understand the implementation process for a blood culture diagnostic stewardship program.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Woods-Hill, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (8):
- United States (8):
  - UCLA Mattel Children's Hospital, Los Angeles, California
  - UCSF Benioff Children's Hospital Mission Bay, San Francisco, California
  - Nemours / AI DuPont Hospital for Children, Wilmington, Delaware
  - Riley Hospital for Children, Indianapolis, Indiana
  - Norton Children's Hospital, Louisville, Kentucky
  - Kravis Children's Hospital, New York, New York
  - New York-Presbyterian Morgan Stanley Children's Hospital, New York, New York
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers. Summary level data will be published.